CLINICAL TRIAL: NCT05658445
Title: Potential Role of microRNA 410 and BIRC7 Pathways in Recurrent Spontaneous Miscarriage
Acronym: microRNA410
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nesma Gamal, faculty of medicine Assuit university, Assiut University
Other Study IDs: As
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2023-12

CONDITIONS: Abortion, Habitual
Keywords: RSA
MeSH Terms: conditions — Abortion, Habitual | interventions — Emergency Shelter

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Months
Biospecimen Retention: Samples With DNA — placental samples (4×6 cm) will be collected from women with miscarriage. Placental tissue from healthy controls (females with normal or caesarean labour)will also be collected. Tissue samples will be removed from the central region of the placenta and processed within 30 min. All samples will be repeatedly rinsed with cold phosphate buffered saline (PBS), and maintained at -80 °C until genetic study of miR-410-5p expression, Integrin alpha-6gene expression and Baculoviral IAP Repeat Containing 7(BIRC7) expression by qRTPCR.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: Female with recurrent unexplained abortion
  Interventions: Other: evacuation
- control: female with normal labour
  Interventions: Other: evacuation

INTERVENTIONS:
Other: evacuation — after complete evacuation of uterus follow abortion

SUMMARY:
The definition of recurrent spontaneous abortion (RSA) has changed over the years, and most societies now advocate defining RSA as two or three consecutive or discontinuous miscarriages with the same sexual partner before 24 weeks gestation

In recent years, the incidence of this disease has been on the rise, occurring in about 1%- 5% of pregnancy in women at childbearing age, and the success rate of second pregnancy in RSA females has been significantly reduced The etiology of RSA is extremely complex, including anatomical factors, genetic factors, endocrine factors, infectious and immune factors, and pre-thrombosis etiology.

However, the cause of the disease is unclear in half of patients and known as unexplained recurrent spontaneous abortion (URSA)

DETAILED DESCRIPTION:
* MicroRNA (miRNA) is a kind of non-coding single-stranded RNA molecule encoded by endogenous genes with a length of about 22 nucleotides . MiRNA negatively regulates gene expression mainly by binding to the 3 'untranslated region (3' UTR) of target mRNA to degrade the target mRNA or inhibit its translation . In recent years, there have been numerous reports about miRNA's involvement in the pathogenesis of RSA, and many of them have focused on how miRNA regulates trophoblast function.
* Additionally, microRNA (miR)-410-5p has been discovered to serve as oncogenes and tumor suppressors altering cell functions in numerous ways including proliferation, apoptosis, biochemistry metabolism, and inflammatory responses in different human malignancies, such as liver cancer, pancreatic cancer, colon cancer, and non-small cell lung cancer. Recent studies showed that miR-410-5p may be involved in the non-cancerous disorder processes such as RSA . Overexpression of miR-410-5p in trophoblast cells inhibited the polarization of M2 macrophages, while knockdown of miR-410-5p was beneficial to recruitment of trophoblast cell and promoted the polarization of M2 macrophages. Furthermore, MicroRNA (miR)-410-5p was discovered to bind with 3'-UTR of ITGA6 .
* The adhesion molecule integrin alpha-6 (ITGA6, CD49f), a member of the integrin family, is overexpressed in many cancers and enhances cell movement and signal output .
* Down-regulation of ITGA6 changed the biological function of trophoblast cells, inhibited cell proliferation, invasion and migration, and induced apoptosis. ITGA6 may affect the biological functions of trophoblast cells by regulating PI3K/AKT and MAPK signaling pathways. MAPK signaling promote apoptosis through inducing releasing of cytochrome c, which in turn induces further caspase activation (caspase-9 and the effector caspases-3, -6, and -7) .
* Baculoviral IAP Repeat Containing 7(BIRC7) encodes the protein Livin which is a member of the inhibitor of apoptosis protein (IAP) family. Livin consists of a single baculoviral IAP repeat domain (BIR) and a RING domian at the C-terminus. The protein inhibits apoptosis by inhibiting proteolytic activation of capsases.
* Currently, the interaction of BIRC7 and NK cells in endometrium/decidual remains unknown. BIRC7 in decidua cell may possess the ability to prevent NK cells from killing embryonic and extraembryonic cells, decreased level of BIRC7 and increased number of NK cells in the RM group attribute to the occurrence of miscarriage

ELIGIBILITY:
Inclusion Criteria: maternal age is between 20 to 30 years and Gestational age before abortion less than 24 weeks.

Female with unexplained two or three consecutive or discontinuous miscarriages with the same sexual partner

Exclusion Criteria:

1. Female with one miscarriage
2. Female with explained causes of miscarriage
3. Female with cancer
4. Female with chronic illness.
5. Pregnant women above 30

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — only females with URSA
Study Population: Female without cancer or chronic illness that exposed to 2 or 3 consecutive or discontinues abortion
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Define a novel hypothesis that may explain the aetiology of URSA | within 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Bochemistry Department, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Undecided